CLINICAL TRIAL: NCT00194480
Title: Treatment of Acute Hepatitis C Virus Infection in Injection Drug Users With Pegylated Interferon for 24 Weeks
Brief Title: Treatment of Acute Hepatitis C Virus Infection With Pegylated Interferon in Injection Drug Users
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Washington (Other)
Responsible Party: Jag H. Khalsa, Ph.D., NIDA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-16066-1; R21DA016066-01 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-10

CONDITIONS: Substance-Related Disorders; Hepatitis
Keywords: Hepatitis C, peg-Interferon, drug abuse
MeSH Terms: conditions — Substance-Related Disorders; Hepatitis; Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PegInterferon (Experimental): Arm 1: 24 weeks of weekly injections of peginterferon Arm 2: control (no treatment)
  Interventions: Drug: Pegylated Interferon

INTERVENTIONS:
Drug: Pegylated Interferon — Weekly injections of pegIntereferon

SUMMARY:
Injection drug use accounts for transmission of a high proportion of Hepatitis C Virus (HCV) infections. The purpose of this trial is to investigate the effectiveness of pegylated interferon in treating injection drug users (IDUs) with acute HCV.

DETAILED DESCRIPTION:
IDUs are at high risk for developing HCV. Pegylated interferon is a man-made form of interferon, a chemical naturally produced by the body that works to fight viruses. Interferon helps to stop HCV from replicating, and helps the immune system to kill HCV. The purpose of this trial is to determine the effectiveness of pegylated interferon in IDUs with HCV.

This trial will last 24 weeks. Participants will be randomly assigned to one of two groups. Group 1 will receive pegylated interferon while group 2 will receive an active control. Injection with either pegylated interferon or control will occur weekly. During each injection visit, participants will be asked about adverse events, including common side effects to interferon such as injection site reactions, headache, myalgias, arthralgias, insomnia, and hair loss. At Weeks 2, 4, and then every 4 weeks thereafter, participants will complete depression self-reports. Laboratory assessments will occur at Week 2, and then on a monthly basis for the remainder of the study. Follow-up assessments will occur every 4 weeks after Week 24.

ELIGIBILITY:
Inclusion Criteria:

* Documented HCV antibody seroconversion within the 12 months prior to study entry
* Serum positive for HCV
* Meets hematologic, biochemical, and serologic criteria at entry visit
* Thyroid stimulating hormone within normal limits
* Hepatitis B surface antigen negative
* Reads at an eighth grade reading level
* Willing to use adequate contraception for the duration of the study
* Plans to remain in the study area for 12 months

Exclusion Criteria:

* Positive test for Hepatitis A antibodies, Hepatitis B antibodies, or HIV antibodies
* Suspected hypersensitivity to pegylated interferon
* Liver disease
* Hemoglobinopathies
* Immune mediated disease
* Significant cardiac or pulmonary disease
* Uncontrolled seizure disorder
* Renal insufficiency with serum creatinine levels greater than 11.5 mb/ml or less than 60 mb/ml
* History of thyroid disease
* Active gout
* Any medical condition requiring or likely to require steroids during the course of study
* Untreated severe psychiatric disorder, as determined by study psychiatrist
* Any condition, which in the opinion of the investigator, would preclude successful completion of the study
* Pregnant or breastfeeding

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-04; Primary Completion 2006-12 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Sustained viral response rate in treatment group versus control (measured at Week 24) | 24 weeks

SECONDARY OUTCOMES:
Adherence rate in the treatment group (measured at Week 24) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chia Wang, MD, MS, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, 325 Ninth Ave 1EC32, Seattle, Washington, United States